CLINICAL TRIAL: NCT02740829
Title: Evaluation of the Effects of Intranasal Glucagon on Endogenous Glucose Production in Humans
Brief Title: Assessment of Intranasal Glucagon on Endogenous Glucose Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 14-8171-A
Record Dates: First submitted 2016-03-08; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: Intranasal placebo
- Intranasal glucagon (Experimental): active intervention
  Interventions: Drug: Intranasal glucagon

INTERVENTIONS:
Drug: Intranasal glucagon — Glucagon will be administered via a nasal dispenser
  Arms: Intranasal glucagon
Drug: Intranasal placebo — Placebo
  Arms: Intranasal placebo

SUMMARY:
Peripheral glucagon action increases hepatic glucose production. In rodents hypothalamic action of glucagon paradoxically suppresses glucose production. Intranasally administered peptides have been shown to preferentially enter the central nervous system. We assessed the effects of intranasal glucagon on hepatic glucose production

DETAILED DESCRIPTION:
Fifteen healthy, lean, non-diabetic males and females will undergo two studies each (single blinded crossover), in random order, 4-6 weeks apart.

Study A. Intranasal placebo administration with measurement of endogenous glucose production under pancreatic clamp conditions.

Study B. Intranasal glucagon (glucagon, Eli Lilly, Canada) administration with measurement of endogenous glucose production under pancreatic clamp conditions Each study participant will be admitted to the Metabolic Test Centre of the Toronto General Hospital the day before the study at 12pm. They will be provided with a standardized dinner (consisting of 7 Kcal/kg; 50% carbohydrate, 30% fat, and 20% protein) and will then be required to fast for 12 hr overnight (can have water but no other food or drinks).

At 7am (t=0) the next day, we will begin a primed, constant intravenous infusion of [6,6-2H2]glucose (D2 glucose; Cambridge Isotope Laboratories, MA; a stable isotope of glucose, the enrichment of which can be measured by GC/MS, allowing us to calculate endogenous glucose production rates). The infusion will continue for 8 hours.

At the same time (7am) a pancreatic clamp will be started for 8 hours in order to suppress pancreatic hormone secretion with somatostatin while providing basal infusions of pancreatic hormones and growth hormone by intravenous infusion. This method will permit us to study the effect of intranasal glucagon on hepatic glucose and TRL production without the confounding effects it may have on pancreatic hormone secretion. A simultaneous infusion of somatostatin (Sandostatin, Novartis Pharma, Miss, ON 30mcg/hr), insulin (Humulin R, Eli Lilly, Scarborough, ON, 0.05mU/kg/min), glucagon (Eli Lilly, Miss, ON 0.325ng/kg/min) and growth hormone (Humatrope, Eli Lilly, Mississauga, ON 3ng/kg/min) will be started and continued throughout the study. All hormones were diluted in 1 liter of normal saline and infused with a syringe pump (B. Braun Medical Inc., Bethlehem, PA). Autologous serum (3 mL), freshly prepared from the subject's blood, was added to the saline as carrier prior to hormone dilution.

A study nurse and/or doctor will be by the bedside throughout the clamp and will be monitoring the participant's blood glucose every 30 minutes after the onset of the clamp and every 10 minutes after administration of glucagon (if clinically indicated, sampling may be more frequent) to ensure participants do not develop hypo/hyperglycemia. Blood samples will be analysed with a glucometer for instant blood glucose readings. If intranasal glucagon reduces endogenous glucose production, a reduction in plasma glucose is likely. 20% dextrose will be administered if necessary to maintain euglycemia At 9 am (+120 minutes) intranasal placebo or glucagon will be administered. The glucagon (Eli Lily, Canada) and placebo (diluent) will be transferred to a metered nasal device (Pharmasystems, Markham, Ontario UPC: 063636 802721, Item 10271) immediately prior to use. This device dispenses 0.1ml (0.1mg) per puff. A maximum of 15 X0.1 ml puffs/vials (7 in 1 nostril and 8 in the other nostril) will be administered at rate of 2 (one in each nostril) every 60 seconds. This dose may be titrated down if necessary to reduce peripheral spillover.

Blood samples will be collected every 30 minutes after the start of the clamp and every 10 minutes after administration of intranasal glucagon or placebo (total of 400 ml). The blood samples will be collected into chilled sterile tubes containing 0.1% EDTA and preservative ( aprotinin, sodium azide) and processed as indicated below.

In order to match peripheral glucagon concentrations between study visits, a small dose of glucagon will likely need to be administered intravenously at 9am, during the placebo arm of the study. Based on the pharmacokinetics of glucagon, we are likely to administer 0.00625mg-0.025mg, although further dose titration may be necessary (maximum dose 0.1mg). Free fatty acids, triglycerides, insulin, glucagon, C-peptide, glucagon-like peptide-1 (GLP-1) and GIP,as well as glucose isotopic enrichment will be measured.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women, aged 18 to 60 years 2. Body mass index 20 to 27 kg/m2 3. Hemoglobin in the normal range. 4. Normal glucose tolerance in response to a 75gram glucose

Exclusion Criteria:

* 1. Study participant with a history of hepatitis/hepatic disease that has been active within the previous two years.

  2. Any current or previous history of biliary disease (including gall stones, biliary atresia and cholecystitis) or pancreatitis.

  3. Any current or previous history of endocrine disease, dyslipidemia or malignancy 4. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal, genitourinary, hematological systems, or has severe uncontrolled treated or untreated hyper/ hypotension (sitting diastolic > 100 or systolic > 180 or systolic<100) or proliferative retinopathy 5. Use of immunosuppressive agents at any time during the study 6. Allergy to any study medication 7. Pregnancy or breastfeeding 8. Heavy smoker 9. Fasting blood glucose > 6.0 mmol/l or known diabetes. 10. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.

  11. Any nasal pathology. 12. Abnormal liver and thyroid function 13. Current addiction to alcohol or substances of abuse as determined by the investigator or of any mental illness.

  14. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation 15. Taking any regular prescription or non-prescription medications at the time of the study. Occasional use of medications such as acetoaminophen or Tylenol 1 or any use of natural health products may be permitted at the discretion of the investigator.

  16. Will not donate blood three months prior to and three months post study procedures

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Endogenous glucose production following intranasal glucagon compared to placebo | 6 hours
  Stable isotope infusion (D2 glucose) will enable assessment of endogenous glucose production by measuring glucose enrichment in plasma by gas chromatogaphy mass spectrometry. During steady state, rate of glucose appearance (Ra) = rate of glucose disappearance (Rd), where Ra = tracer infusion rate /plasma tracer enrichment. Endogenous glucose production (EGP) rate = Ra - glucose infusion rate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dash S, Xiao C, Stahel P, Koulajian K, Giacca A, Lewis GF. Evaluation of the specific effects of intranasal glucagon on glucose production and lipid concentration in healthy men during a pancreatic clamp. Diabetes Obes Metab. 2018 Feb;20(2):328-334. doi: 10.1111/dom.13069. Epub 2017 Sep 14. PMID 28730676